CLINICAL TRIAL: NCT00193778
Title: A Randomized Trial To Assess The Impact Of Loco-Regional Treatment On Survival Of Patients With Metastatic Breast Cancer At First Presentation
Brief Title: Assessing Impact of Loco-regional Treatment on Survival in Metastatic Breast Cancer at Presentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH/153/2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cancer of the Breast
Keywords: Metastatic breast cancer; Locoregional treatment; Survival
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loco Regional Treatment Arm (LRT) (Experimental): Surgery for breast cancer. (MRM/BCT)
  Interventions: Procedure: Surgery for breast cancer
- No Loco-regional Treatment Arm (Active Comparator): No surgery for Breast cancer
  Interventions: Other: No Loco-regional treatment

INTERVENTIONS:
Procedure: Surgery for breast cancer — This group will receive standard loco-regional treatment i.e. surgery (modified radical mastectomy (MRM)/ Simple SMAC/BCT) +/- radiotherapy
  Arms: Loco Regional Treatment Arm (LRT)
Other: No Loco-regional treatment — This group will not receive any loco-regional treatment
  Arms: No Loco-regional Treatment Arm

SUMMARY:
Traditionally metastatic breast cancer patients are not offered loco-regional treatment except in cases of fungation or bleeding. However, scientific evidence for such omission of loco-regional treatment in metastatic breast cancer patients is lacking. On one hand, studies have shown that removal of primary tumor at times leads to complete disappearance of metastases and improvement in survival in renal cell carcinoma patients. However, such studies have never been performed in other solid tumors. On the other hand, there is a strong body of evidence in experimental settings that show that removal of primary tumor allows growth of metastasis. There is lack of similar data in humans in clinical settings. Offering loco-regional treatment in metastatic breast cancer patients in a setting of randomized controlled trial will help in improving survival of such patients and understanding the natural history of breast cancer.

DETAILED DESCRIPTION:
PRESENT KNOWLEDGE:

Loco-regional treatment should not be attempted in metastatic breast cancer patients is a traditional teaching, which lacks scientific basis. Omission of loco-regional treatment can not be part of standard care if the scientific evidence is inadequate. Today such a treatment is offered for fungation and/or bleeding.

Studies in metastatic renal cell carcinoma have shown that removal of primary tumor can cause disappearance of metastases [1] and improve survival[2,3]. The exact mechanism of this phenomenon is not understood. Although immunologic mechanisms have been suggested, these remain largely unproven.[1] On the contrary, metastases autonomy hypothesis on animal models suggests that removal of primary tumor renders autonomy to metastases, which start growing rapidly.[4] The suggested mechanism for this is anti-angiogenic/ angiostatic activity of the primary tumor. However, such studies have never been performed in human subjects.

Which hypothesis is true? What does removal of primary tumor cause - suppression or stimulation of growth of metastases? Whether such suppression or stimulation affects survival? These are few questions, which need to be answered to improve our understanding of natural history of breast cancer. vascular endothelial growth factor (VEGF)[5], basic fibroblast growth factor (bFGF)[6] are some of the angiogenic and proliferative factors which stimulate tumor/ metastasis growth. Angiostatin[7] and Endostatin[8] are the some of the inhibitors of angiogenesis. It is the balance between angiogenic factors and anti-angiogenic factors that determines the tumor/metastases growth[7]. Lot of ongoing research[9] is focused on administration of Angiostatin and Endostatin to tilt this balance in favor of anti-angiogenesis. Does removal of the primary tumor change this balance? And what impact this change in balance (if any) have on survival? These questions have not been answered by in-vivo studies in humans. Demonstration of such effects or absence of these effects can help us in refining our therapeutic targets in metastatic patients.

There is dearth of reliable data on change in the levels of angiogenic, proliferative growth factors and anti-angiogenic factors in relation to the time after removal of primary. Removal of primary tumor resulted in growth of metastases in animal experiments in five days[4] and the metastases tripled in size by thirteenth day. Hence, we decide to measure levels of these factors at the end of one week following surgery and at the end of three months.

This study aims at:

Firstly, assessing impact of loco-regional treatment on survival in metastatic breast cancer patients.

Secondly, understanding the mechanism of suppression/ stimulation of growth of the metastases through measurement of angiogenic, proliferative growth factors and anti-angiogenic factors before and after intervention.

TRIAL DESIGN:

Patients with metastatic breast cancer diagnosed by incision biopsy and staging investigations will undergo six cycles of anthracycline-based chemotherapy. At the end of chemotherapy, these patients will be randomized into two groups. First group will receive standard loco-regional treatment i.e. surgery (modified radical mastectomy(MRM)/ Simple Mastectomy with Axillary Clearance (SMAC)/ Breast Conservation Therapy (BCT) +/- radiotherapy (depending on type of surgery performed or histopathology report). Second group will not receive any loco-regional treatment.

INVESTIGATIONS:

A. Diagnostic: Incision biopsy for primary diagnosis and estrogen receptor (ER)/ progesterone receptor (PgR) status.

B. Staging:

* Liver function tests
* Chest X-ray & USG - Abdomen & pelvis &/ CECT chest with Upper Abdomen
* Bone scan with relevant x-ray skeletal survey (MRI in doubtful cases)

ELIGIBILITY:

Inclusion criteria:

1. Metastatic breast cancer patients with expected survival of at least one year
2. Age 21-65 years

Exclusion criteria:

1. Patients who are not fit to receive anthracycline based chemotherapy.
2. More than two visceral organ involvement.
3. Multiple liver metastases with deranged liver function tests serum glutamic oxaloacetic transaminase (SGOT) / serum glutamic-pyruvic transaminase (SGPT) more than four times the upper normal limit).
4. Locally static or progressive disease or systemically progressive disease as shown by repeat staging investigations guided by worsening symptoms.
5. Ulceration/ fungation/ bleeding after completion of chemotherapy, which mandates surgery.
6. Expected survival of less than six months after completion of chemotherapy.
7. Unfit for anesthesia due to metastatic disease.

CONSENT AND RANDOMIZATION:

Computerized randomization will be carried out at the central office after confirmation of eligibility and obtaining informed written consent. Randomization will be stratified by

1. Visceral or bone and/ or soft tissue metastasis.
2. Less than or equal to 3, or more than three metastases.
3. Hormone responsive or non-responsive tumor.

TRIAL SIZE AND ACCRUAL:

Breast cancer patients who have metastatic disease at presentation have a median survival of eighteen months. Detection of six-month improvement in this survival with 95% confidence and 80% power by a two tailed analysis will require a minimum of 350 patients.

METHODOLOGY:

1. All eligible patients will be provisionally marked for the trial.
2. Number and sites of all the metastases will be documented along with the size.
3. Patients will receive maximum of six cycles of Cyclophosphamide (600 mg/m2), Adriamycin (60 mg/m2), 5- Fluoro-Uracil (600 mg/m2).
4. Patients will be reassessed at the end of chemotherapy (approximately five months later). Staging investigations viz. CECT thorax and upper abdomen (in cases of visceral metastasis) and relevant X-rays will be repeated. All eligible patients will be randomized into two groups (stratified randomization). First group will undergo standard loco-regional treatment (surgery followed by radiotherapy depending on histopathology report or type of surgery performed e.g. BCT) and surgical oophorectomy (at the time of surgery) followed by hormone therapy (in ER and/ or PgR positive pre-menopausal patients). Postmenopausal patients will receive hormone therapy. Second group will be started on hormone therapy (all ER and/ or PgR positive and/ or postmenopausal patients). Hormone therapy will be in the form of Aromatase inhibitors (Letrozole 2.5mg OD/ Anastrozole 1.0mg OD)
5. All patients in loco-regional treatment group will have two or three blood samples (10-cc blood in plain bulbs) collected. These samples will be used for estimation of VEGF, bFGF, Angiostatin and Endostatin by ELISA.

   Sample 1: A day prior to surgery. Sample 2: Seventh post operative day. Sample 3: Three months after the surgery.
6. The metastases will be reassessed after twelve weeks of surgery for any change in size and number by repeat staging investigations viz. CECT thorax and upper abdomen (in cases of visceral metastasis) and relevant X-rays and again on symptomatic progression.

Patients with symptomatic bony metastases will in addition receive local radiotherapy (wherever indicated) and/ or bisphosphonates (wherever indicated).

Patients in both the arms will undergo metastasectomy wherever indicated.

PATHOLOGY: Pathological tumor size, number of axillary lymph nodes dissected and number positive for metastasis, histological type of the primary tumour (infiltrating duct carcinoma with standard grades, infiltrating lobular carcinoma, other rare histologies[medullary, papillary, colloid etc.]), presence or absence of lymphatic, vascular and peri-neural invasion should be noted in all patients. Estimation of other biological markers ER, PgR is mandatory. Entries will be made in case report forms (CRFs).

END POINT:

Primary: 1. Overall survival (time to death) 2. Progression free survival

Secondary:

Changes in VEGF, bFGF, Angiostatin and Endostatin.

DATA COLLECTION, QUALITY CONTROL AND ANALYSIS:

Data collection will be carried out by individual clinician on prescribed forms: Pre-randomization form, primary data sheet, and pathology information. At least 20% of the data will be cross-checked by internal/external review. The trial centre data manager with the help of individual clinician will maintain completeness of data but the latter will be responsible for the correctness of information. All forms will be maintained in duplicate at the central trial office.

Data monitoring committee will periodically review the trial. Univariate comparison between randomization arms will be carried out using chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer at first presentation with an expected survival of at least one year

Exclusion Criteria:

1. Patients who are not fit to receive anthracycline based chemotherapy.
2. More than two visceral organ involvement.
3. Multiple liver metastases with deranged liver function tests (SGOT/SGPT more than four times the upper normal limit).
4. Locally static or progressive disease or systemically progressive disease as shown by repeat staging investigations guided by worsening symptoms.
5. Ulceration/ fungation/ bleeding after completion of chemotherapy, which mandates surgery.
6. Expected survival of less than six months after completion of chemotherapy.
7. Unfit for anaesthesia due to metastatic disease.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2005-02; Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival (OS) : Time interval between randomization and death
Progression free survival | 3 years
  PFS: Time interval between randomization and first date of progression of disease

SECONDARY OUTCOMES:
Changes in VEGF, bFGF, Angiostatin and Endostatin | 5 years
  The secondary endpoints include the assess of loco-regional treatment on levels

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, MS (Surgery), Principal Investigator — Tata Memorial Hospital, Ernest Borges Road, Parel, Mumbai 400 012
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Lokich J. Spontaneous regression of metastatic renal cancer. Case report and literature review. Am J Clin Oncol. 1997 Aug;20(4):416-8. doi: 10.1097/00000421-199708000-00020. PMID 9256902
- [Background] Flanigan RC, Salmon SE, Blumenstein BA, Bearman SI, Roy V, McGrath PC, Caton JR Jr, Munshi N, Crawford ED. Nephrectomy followed by interferon alfa-2b compared with interferon alfa-2b alone for metastatic renal-cell cancer. N Engl J Med. 2001 Dec 6;345(23):1655-9. doi: 10.1056/NEJMoa003013. PMID 11759643
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Fisher B, Gunduz N, Coyle J, Rudock C, Saffer E. Presence of a growth-stimulating factor in serum following primary tumor removal in mice. Cancer Res. 1989 Apr 15;49(8):1996-2001. PMID 2702641
- [Background] Kim KJ, Li B, Winer J, Armanini M, Gillett N, Phillips HS, Ferrara N. Inhibition of vascular endothelial growth factor-induced angiogenesis suppresses tumour growth in vivo. Nature. 1993 Apr 29;362(6423):841-4. doi: 10.1038/362841a0. PMID 7683111
- [Background] Hori A, Sasada R, Matsutani E, Naito K, Sakura Y, Fujita T, Kozai Y. Suppression of solid tumor growth by immunoneutralizing monoclonal antibody against human basic fibroblast growth factor. Cancer Res. 1991 Nov 15;51(22):6180-4. PMID 1718597
- [Background] O'Reilly MS, Holmgren L, Shing Y, Chen C, Rosenthal RA, Moses M, Lane WS, Cao Y, Sage EH, Folkman J. Angiostatin: a novel angiogenesis inhibitor that mediates the suppression of metastases by a Lewis lung carcinoma. Cell. 1994 Oct 21;79(2):315-28. doi: 10.1016/0092-8674(94)90200-3. PMID 7525077
- [Background] O'Reilly MS, Holmgren L, Shing Y, Chen C, Rosenthal RA, Cao Y, Moses M, Lane WS, Sage EH, Folkman J. Angiostatin: a circulating endothelial cell inhibitor that suppresses angiogenesis and tumor growth. Cold Spring Harb Symp Quant Biol. 1994;59:471-82. doi: 10.1101/sqb.1994.059.01.052. No abstract available. PMID 7587101
- [Derived] Badwe R, Hawaldar R, Nair N, Kaushik R, Parmar V, Siddique S, Budrukkar A, Mittra I, Gupta S. Locoregional treatment versus no treatment of the primary tumour in metastatic breast cancer: an open-label randomised controlled trial. Lancet Oncol. 2015 Oct;16(13):1380-8. doi: 10.1016/S1470-2045(15)00135-7. Epub 2015 Sep 9. PMID 26363985